CLINICAL TRIAL: NCT06074094
Title: Effect of Probiotic Supplementation on Non-alcoholic Fatty Liver Disease in Patients Attending Family Medicine Clinic in Ain Shams University Hospitals
Brief Title: Probiotic Supplementation IN NAFLD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: probiotic and NAFLD
Record Dates: First submitted 2023-09-13; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-06

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiotic group (Experimental): Healthy lifestyle habits and standard diet was recommended for participants ,Probiotic supplementation (Lacteol fort 10 billion) which contains culture medium and lactobacillus LS as active ingredients was administered in the form of oral sachets once daily for 12 weeks.
  Interventions: Drug: Control Test
- standard treatment group (Active Comparator): Healthy lifestyle habits and standard diet was recommended for participants ,
  Interventions: Drug: Control Test

INTERVENTIONS:
Drug: Control Test — Lacteol fort 10 billion which contains culture medium and lactobacillus LS as active ingredients
  Other Names: standard treatment group

SUMMARY:
this study aimed to evaluate the effectiveness of Probiotics supplementation (lactobacillus) on NAFLD fibrosis score.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a disease characterized by accumulation of fat (> 5% of the liver tissue), in the absence of alcohol abuse or other chronic liver diseases. NAFLD can cause liver inflammation and progress to non-alcoholic steatohepatitis (NASH), fibrosis, cirrhosis or hepatocellular carcinoma (HCC).

The global prevalence of NAFLD in adults is estimated to be approximately 25%.The prevalence of NAFLD increases with increasing body mass index. in 2012 Chalasani et al, reported that 67% of overweight and 94% of obese individuals have NAFLD.

There is a consensus regarding increasing worldwide prevalence of NAFLD and its impact on health, especially the progression to liver cirrhosis and hepatocellular carcinoma. Longitudinal studies of NAFLD have reported an increase in all-cause mortality, cardiovascular mortality, and liver-related mortality , NAFLD carries a large economic burden and therefore poor health-related quality of life.

Lifestyle changes (diet and exercise) are the major and first suggestions of the guidelines ,as regard pharmaceutical interventions, agents with potential benefit in NASH include thiazolidinediones (TZDs), statins although they are well recognized in the treatment of dyslipidemia, their use as a specific treatment for NAFLD is not well evidenced.

There is some data suggest that disruptions in the gut microbiome may play a role in the pathogenesis of NAFLD and progressions to NASH.

A probiotic is a live microbial culture or cultured dairy product, which plays an important role in health. Probiotics for the treatment of NAFLD are seemingly a promising treatment option. Relatively easy availability, low cost, and absence of serious side effects make probiotics a lucrative choice.

liver biopsy remains the gold standard for NAFLD diagnosis but it is impractical as a diagnostic tool because it is invasive and expensive.

NAFLD fibrosis score constructed from routine clinical and laboratory variables can accurately predict the presence or absence of advanced fibrosis in NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age between18 and 60
* BMI ≥ 25 kg/m2
* Sonographic findings of NAFLD +/- elevated liver enzymes (not more than 2 folds increase).

Exclusion Criteria:

* ▪ Any evidence of chronic liver diseases including viral hepatitis (B and C), auto immune hepatitis.

  * History of alcohol drinking.
  * Chronic medication use (drugs that cause elevated liver enzymes, recent antibiotic use or paracetamol use in the last month)
  * Persistent elevation of liver enzymes for 3 months.
  * History of DM.
  * History of statin therapy for cardiovascular disease (CVD).
  * History of recent operation.
  * History of gastroenteritis or diarrhea in the last 2 week.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
non alcoholic fatty liver disease (NAFLD) fibrosis score | 12 week of probiotic supplementation
  NAFLD fibrosis score constructed from routine clinical and laboratory variables can accurately predict the presence or absence of advanced fibrosis in NAFLD This scoring system had an area under the ROC curve of 0.88 (95% CI 0.85-0.92). 2 cutoff points were selected to identify the presence (> 0.676) and absence (< -1.455) of significant fibrosis.

SECONDARY OUTCOMES:
ALT , AST | 12 week of probiotic supplementation
  effect of probiotic on ALT and AST
body mass index (BMI) | 12 week of probiotic supplementation
  effect of probiotic on body mass index (BMI)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
when appropriate.

REFERENCES:
- [Derived] Abd El Hamid AA, Mohamed AE, Mohamed MS, Amin GEE, Elessawy HAA, Allam MF. The effect of probiotic supplementation on non-alcoholic fatty liver disease (NAFLD) fibrosis score in patients attending a tertiary hospital clinic in Cairo, Egypt. BMC Gastroenterol. 2024 Oct 8;24(1):354. doi: 10.1186/s12876-024-03424-3. PMID 39379797
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28521870/
- See also: Related Info — https://www.nice.org.uk/guidance/ng49